CLINICAL TRIAL: NCT02693808
Title: New Treatment for Patients With Temporal Hollowing After Lateral Wall Decompression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/1175
Record Dates: First submitted 2015-12-04; First posted 2016-02-29 (Estimated); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Thyroid-Associated Ophthalmopathy
Keywords: Temporal hollowing; Lateral orbital wall decompression; Thyroid eye disease
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous fat injection (Active Comparator): Patients have undergone lateral orbital wall decompression on both sides. Temporal hollowing after surgery will be treated with injection on one side with autologous fat and the other side with long-lasting hyaluronic acid.
  Interventions: Procedure: Autologous fat injection; Procedure: Hyaluronic acid injection
- Hyaluronic acid injection (Active Comparator): Patients have undergone lateral orbital wall decompression on both sides. Temporal hollowing after surgery will be treated with injection on one side with autologous fat and the other side with long-lasting hyaluronic acid.
  Interventions: Procedure: Autologous fat injection; Procedure: Hyaluronic acid injection

INTERVENTIONS:
Procedure: Autologous fat injection — Injection in one side with autologous fat and the other side with hyaluronic acid.
Procedure: Hyaluronic acid injection — Injection in one side with autologous fat and the other side with hyaluronic acid.

SUMMARY:
The purpose of this study is to determine whether injection of autologous fat or hyaluronic-acid injections in temporal region are effective in the treatment of temporal hollowing after lateral wall decompression in patients with thyroid eye disease.

DETAILED DESCRIPTION:
Grave's disease is one of the most common autoimmune diseases. Thyroid eye disease is affecting nearly 50% of patients with Grave's disease. Surgical treatment may address several of the manifestations, including the increased volume of the orbital contents. Decompression of the orbit can be achieved by removing the lateral orbital walls; "lateral wall decompression".

In a retrospective study at the Department of Ophthalmology, Haukeland University Hospital, about half of the patients had a disfiguring hollowing in the temporal region after lateral wall decompression. The patient reported outcome of the procedure is clearly an indication for further esthetic treatment. However, until now the treatment option for these patients have been limited, or simply neglected. The investigators have contacted over 40 patients with this complication that want treatment.

In this project the investigators will treat bilateral hollowing with injection of autologous fat in one temporal region and hyaluronic-acid injections on the opposite side. Participants with unilateral hollowing will be randomized to one of the treatment options. Outcomes will be evaluated by clinical examination, photographs and ultrasound volume measurement at 6, 12, 18 and 24 months postoperatively. The participants will be retreated at these follow up intervals if necessary.

The project will be an interventional, prospective follow-up study and is approved by the regional ethics committee. The study will be the first of its kind to date as the investigators will be able to prospectively evaluate the effect of autologous fat injections to hyaluronic-acid injections in the same patient for the same condition.

ELIGIBILITY:
Inclusion Criteria:

* Disfiguring temporal hollowing after lateral wall decompression.
* The participant want treatment for temporal hollowing

Exclusion Critera:

* The participant dont want treatment for temporal hollowing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with satisfactory objective cosmetic and functional outcome | 2 years
  Evaluation of photographs (1 to 3/Normalized to disfiguring)

SECONDARY OUTCOMES:
Volume of injected substance measured by ultrasonography | 2 years
  ml
Number and type of complications | 2 years
  Hematoma, infection, embolization.
Number of reinjections | 2 years
  Number.
Number of patients with satisfactory subjective cosmetic and functional | 2 years
  Patient reported perception of outcome (1 to 3/Normalized to disfiguring)

CONTACTS AND LOCATIONS:
Overall Officials: Eyvind Rødahl, MD PhD, Principal Investigator — University of Bergen
Locations (1):
- Department of Ophthalmology Haukeland University Hospital, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McNichols CH, Hatef DA, Cole P, Hollier LH, Thornton JF. Contemporary techniques for the correction of temporal hollowing: augmentation temporoplasty with the classic dermal fat graft. J Craniofac Surg. 2012 May;23(3):e234-8. doi: 10.1097/SCS.0b013e31824de5b8. PMID 22627443
- [Result] Ueland HO, Nilsen RM, Rodahl E, Jensen SA. Hyaluronic acid is superior to autologous fat for treatment of temporal hollowing after lateral orbital wall decompression: A prospective interventional trial. J Plast Reconstr Aesthet Surg. 2019 Jun;72(6):973-981. doi: 10.1016/j.bjps.2018.12.031. Epub 2018 Dec 14. PMID 30679116